CLINICAL TRIAL: NCT06820034
Title: Empowering Smoking Cessation for People With High Levels of Stress and Low Social Support in Oklahoma and the ACS South Region
Brief Title: Empowering Cessation ACS South Region
Acronym: CHERC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17874; 1181502 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-01-28; First posted 2025-02-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
Keywords: smoking cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation support + volunteering (Experimental): This group will receive remotely-delivered smoking cessation support by using the National Cancer Institute's smoking cessation app and receive combination nicotine replacement therapy (NRT; i.e., lozenges/gum, patches). Additionally, they will engage in sexual and/or gender minority (SGM)-serving online volunteer activities (≥4 sessions) and a digital hub to foster interaction across Oklahoma, Texas, and Arkansas.
  Interventions: Other: Empowering Cessation for the ACS South
- Smoking cessation support ONLY (No Intervention): Participants in this group will receive remotely-delivered smoking cessation support by using the National Cancer Institute's smoking cessation app and receive combination nicotine replacement therapy (NRT; i.e., lozenges/gum, patches).

INTERVENTIONS:
Other: Empowering Cessation for the ACS South — All participants (N=400) will receive remotely-delivered smoking cessation support comprised of the National Cancer Institute's (NCI) free smoking cessation app and 12 weeks of mailed over-the-counter NRT (nicotine patches, gum or lozenges).. While receiving smoking cessation support, participants in the intervention group (n=200) will also engage in SGM-serving online volunteer activities (≥4 weekly sessions lasting ~1.5 hours each), the protocols for which will be developed in Phase 1 to address the needs of OK, AR, and TX communities. Volunteer sessions will be facilitated by an SGM culturally-competent facilitator employed by the research team (i.e., community partner organizations will not run volunteer sessions). The intervention group will also be added to a digital hub (i.e., a private Reddit group) for 12 weeks to foster social support and exchange of ideas between participants/community partners across the three states.
  Arms: Smoking cessation support + volunteering

SUMMARY:
Sexual and/or gender minority (SGM) people face a disproportionate burden of cancer risk, and tobacco use is a key modifiable risk factor. SGM tobacco-related disparities are especially pronounced in places with high levels of stigma against SGM people. This community-engaged and remotely-delivered Research Scholar Grant project will evaluate an empowerment-based smoking cessation intervention tailored for SGM people in high-stigma places. In partnership with Freedom Oklahoma (OK) and a Community Advisory Board from Arkansas (AR) and Texas (TX) this projects aims to: (1) Adapt SGM-serving volunteer activities from the Oklahoma intervention pilot study for delivery in nearby states; (2) Test intervention efficacy among SGM adults in OK, AR, and TX; (3) Identify treatment mechanisms.

ELIGIBILITY:
Exclusion criteria:

* Currently using other smoking cessation treatments.
* Unable or unwilling to use Nicotine Replacement Therapy (NRT)
* Serious psychological distress (i.e., score of 13 ≥ 18 on the Kessler Psychological Distress (PD) Scale-6 19)

Inclusion criteria will be:

1. ≥ 18 years old
2. sexual and/or gender minority-identified (SGM) (see definition below)
3. living in Oklahoma, Texas, or Arkansas (verified by address)
4. a current cigarette smoker (see definition)
5. willing to quit smoking within 30 days of enrollment (see definition)
6. ability to read and speak English 'well' or 'very well'
7. ≥ weekly internet access
8. willing and able to participate in SGM-serving volunteer activities.
9. own a smartphone

Sexual minority identity will be indicated by selecting any non-heterosexual response option(s) from: Heterosexual (Straight); Gay or Lesbian; Bisexual; Something else (please state)." Participants will indicate the sex assigned on their birth certificate (i.e., natal sex). Gender minority identity will be indicated by "Trans male/Trans man;" "Trans female/Trans woman;" "Gender queer/Gender non-conforming;" "Different identity (please state)" or a binary identity (male or female) non-concordant with natal sex.

Current cigarette smoking will be indicated by ≥100 lifetime cigarettes and currently smoking cigarettes "every day" or "some days".

High SGM stigma states are defined as the 22 states wherein ˂60% of the population 'thinks that homosexuality should be accepted'. High SGM stigma municipalities are defined as one of the 246 U.S. municipalities (out of the 496 scored from all U.S. states) that scored below the median (71) on the HRC Municipal Equality Index.

Willingness to quit smoking will be assessed with a single item: "Are you willing to quit smoking cigarettes within 30 days after enrolling in this study? (yes/no)". To be classified as 'ready to quit smoking,' participants will report readiness to quit in the next 30 days and at least 1 past-year quit attempt (i.e., in the "Preparation" stage of change).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically-verified 7-day Point Prevalence Abstinence (PPA) at 26 weeks | 26 weeks post-quit-date
  Self-reported smoking cessation abstinence will be biochemically verified with the iCOQuit Smokerlyzer expired carbon monoxide device 26 weeks after the participant's quit smoking date.

SECONDARY OUTCOMES:
Social Support | Week 0; Week 12
  Patient-Reported Outcomes Measurement Information System (PROMIS) emotional support scale.
  5-point Likert scale; Strongly disagree = least support ... Strongly agree = most support
Smoking intensity | Week 0, Week 12, Week 26
  -Smoking intensity will be assessed by past-week smoking days and past-week cigarettes per smoking day.
  Greater number of smoking days and great number of cigarettes per day = greater smoking intensity
Adaptive coping with minority stress | Week 0; Week 12
  Brief- Coping Orientation to Problems Experienced Inventory (COPE) [adapted]
  5-point Likert scale; Strongly disagree to Strongly agree. Higher score = more coping
Self-efficacy | Week 0, Week 12, Week 26
  -Self-Efficacy Scale/Confidence (SESC) Scale of 10 Very confident to 1 not at all confident. Higher score = greater self-efficacy to quit smoking
Motivation to quit smoking | Week 0, Week 12, Week 26
  -Motivation to change (Stages of Change [SoC] scale) 0 (Not at all ready)-----------------------10 (Extremely ready/already quit) Higher score = more motivation to quit smoking
Internalized transphobia | Week 0; Week 12
  Gender Minority Stress and Resilience: Internalized transphobia subscale 5-point Likert scale; Strongly disagree to Strongly agree Higher score = greater internalized transphobia
Prosociality | Week 0; Week 12
  Well-Being in Prosociality [Chi K, Almeida DM, Charles ST, et al. Daily prosocial activities and well-being: Age moderation in two national studies. Psychology and Aging 2021;36(1):83.] 5-point Likert Scale: Strongly agree to Strongly disagree Higher score indicates greater prosociality
Nicotine Replacement Therapy (NRT) Adherence | Weeks 1, 3, 5, 7, 9, 11
  Medication Adherence Questionnaire (MAQ) Yes=0; No=1; higher score = greater adherence
Smoking cessation app engagement | Weeks 3, 5, 7, 9, 11
  Self-report of number of times per day participant opened app, on average, over the past week. Greater number of times opened = greater engagement
Intervention satisfaction | Weeks 3, 5, 7, 9, 12
  Validated measures of intervention feasibility, acceptability, and appropriateness (Weiner et al, 2017) 5 point ordinal scale from "completely disagree=0" to "completely agree=4"; higher score = greater intervention satisfaction
Sexual Orientation Identity Pride | Week 0, Week 12
  Lesbian, Gay, and Bisexual Identity Scales: Identity Concealment Motivation subscale; Internalized Homonegativity; Identity Acceptance Concerns 6-point scale: 1=Disagree strongly... 6=Strongly agree Higher score = greater identity concerns
Gender identity and expression pride | Week 0, Week 12
  Gender Minority Stress and Resilience: Gender Identity & Expression Pride subscale 5-point Likert scale; Strongly disagree to Strongly agree Higher score = greater gender identity and expression pride

IPD SHARING:
Plan to Share IPD: No